CLINICAL TRIAL: NCT03222180
Title: A Crowdsourced Social Media Portal for Parents of Very Young Children With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Jessica Pierce, Research Scientist, Nemours Children's Clinic
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1DP3DK108198 (NIH)
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: The study design consists of randomization of parents of 150 children with T1D to either Website (n=100) or Usual Care (n=50) for 6 months followed by all participants reverting to the Website condition for the subsequent 6 months.
Who Masked: Outcomes Assessor
Masking Description: Persons administering and scoring study questionnaires will be blinded to the participants' group assignments,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Website (Experimental): Participants will be provided with password-protected access to use of the online resource created during the first phase of the project during the one year randomized controlled trial. Participants' children with T1D will receive Usual Care for T1D as described below.
  Interventions: Behavioral: Website
- Usual Care (No Intervention): Participants' children with T1D will receive care for T1D at their respective institutions equivalent to that received by comparable patients who do not enroll in the trial. At all sites, Usual Care is designed to be consistent with the current American Diabetes Association Standards of Care for T1D in this clinical population.

INTERVENTIONS:
Behavioral: Website — Participants in the Website condition will be provided with password-protected access to the online resource created for this trial that provides a variety of information, support and guidance that could permit them to adapt more effectively to the demands of parenting a very young child with type 1 diabetes.
  Arms: Website

SUMMARY:
The first 2 years of this project consisted of user-centered design and development of an online resource designed by and for parents of very young children with type 1 diabetes (under 6 years old). That phase of the work has been completed and recruitment has begun for the second phase, which is a randomized controlled trial to evaluate the effects of use of this resource on a variety of pertinent child and parent outcomes. INTERESTED, ELIGIBLE PARENTS OR GUARDIANS CAN LEARN MORE BY NAVIGATING TO: www.bit.ly/youngT1D

DETAILED DESCRIPTION:
In response to PA-DK-14-022, the researchers propose to design and test an intervention to improve management of type 1 diabetes (T1D) in very young children (<6 years). Parents of very young children with T1D (YC-T1D) often experience distress and anxiety that can impede T1D care, threatening the child's current and future adaptation to T1D.Typical health care often does not equip parents to contend with these issues, but YC-T1D parents can offer support/guidance to each other to promote parental coping and thus child outcomes. The many obstacles to direct interaction among parents suggest that social media may be an efficacious way to facilitate timely, meaningful and needed social support such as parenting guidance, affective support, provision of information, and sharing of creative solutions to common T1D management problems in YC-T1D. Many good social media resources exist, but there is not a focused portal that facilitates parents' access to these resources, nor have potential benefits been validated empirically. The researchers applied crowdsourcing methods to achieve the iterative development and initial evaluation of an online resource designed by and for YC-T1D parents with continuous input from health professionals and technical expertise in crowdsourcing and application development provided by our web development agency partners (e-city interactive, Philadelphia) and Nemours web development team.

Crowdsourcing is a flexible online activity that has been applied to diverse problems in many fields, including public health, with four elements: 1.) An organization that has a task it needs to be performed, (development of an online resource that meets the needs of parents of YC-T1D); 2.) A community, "the crowd", that agrees to perform the necessary tasks voluntarily (here parents of YC-T1D, T1D clinicians, and professional application developers); 3.) An online environment that allows the work to take place by enabling collaboration between the crowd and the organization, (the infrastructure proposed in this grant); and 4.) Mutual benefit for the organization and members of the crowd (better glycemic control, improved quality of life and decreased burden of care for YC-T1D and their families).

To the researchers' knowledge, crowdsourcing has not been applied to the design and development of online health behavior resources such as that proposed in this application. They will design the portal with stakeholders based on principles of User-Centered Design and then collect preliminary data needed to justify and then conduct a rigorous controlled trial of the effectiveness of an online resource that will provide parents of YC-T1D (<6 years old) with timely, responsible, safe and effective support and guidance regarding parental management of common behavioral, affective and cognitive barriers to effective T1D care in this age group. The proposed work will address these specific aims:

Aim 1 (Completed): The team used crowdsourcing methods to 1.) Identify the most important concerns about management of YC-T1D from key stakeholders (parents, pediatric endocrinologists, diabetes nurses, dietitians, psychologists and social workers) to specify content areas that the online resource should address; 2.) Collaborate with parents (with available input from T1D professionals) to design the optimal content, structure, functions and governance of a social media resource for parents of YC-T1D to improve daily T1D care and problem solving, to enhance parental coping with sources of distress and care burden that uniquely affect this clinical population and to facilitate parents' access to and use of other beneficial resources of the diabetes online community.

Aim 2 (Completed): The researchers iteratively incorporated the knowledge, experience and perspectives gained in Aim 1 to systematically build and refine an online resource enabling parents of very young children with T1D to obtain real-time emotional support, information and parenting guidance, enabling them to cope more effectively with the daily demands of diabetes management in this population. The team relied on the web development agency partners, Nemours web development team, and ongoing stakeholder input.

Aim 3 (Completed): The researchers will conduct a randomized controlled trial of a final version of the online resource with parents of at least 150 children <6 years old who receive T1D care at any Nemours operating entity in the Delaware Valley and Florida or who enroll in response to online announcements. The team will explore treatment effects on metabolic, behavioral and affective outcomes of T1D care, patterns of portal utilization by parents and users' feedback on website use during and after the trial.

Having designed, built, tested, validated and refined the proposed online resource, the team will be well-positioned to plan and complete a rigorous randomized controlled trial to evaluate effects of portal use/access on metabolic, behavioral, affective and social outcomes of T1D care for YC-T1D. While completing Aim 3, the researchers will solidify partnerships with several key organizations (PEDSnet, T1D Exchange, JDRF, American Diabetes Association) to enable economical completion of a major multisite trial. The design of the proposed preliminary RCT will position the team to propose a completely electronic multisite RCT that does not require face to face contact between parents and the research team and can be completed totally in cyberspace.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian of a child with T1D < 6 years old at enrollment
* Child and parent/guardian live in the United States
* Parent is able to read and comprehend written English
* Access to the internet

Exclusion Criteria:

* Inability to read or comprehend study questionnaires or website content

INTERESTED, ELIGIBLE PARENTS OR GUARDIANS CAN LEARN MORE BY NAVIGATING TO: www.bit.ly/youngT1D

Ages: 1 Day to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 174 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Parental adjustment | 12 months
  Questionnaire scores
Child adjustment | 12 months
  Questionnaire scores
Glycated hemoglobin (Hemoglobin A1c) | 12 months
  Change in child's glycated hemoglobin level during the trial

SECONDARY OUTCOMES:
Severe hypoglycemia | 12 months
  Frequency of severe hypoglycemic events
Health care utilization | 12 months
  Hospitalizations or ED visits associated with T1D
Website utilization | 12 months
  Automated collection of website logins, navigation, duration of use, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
After the results pertinent to the specific aims have been accepted for publication, a de-identified data set will be placed in a publicly accessible secure location along with an accompanying data dictionary. Access to the data set will be limited to those persons who sing and submit a data use agreement that ensures protection of the confidentiality of the study participants.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Once the results pertinent to each of the specific aims have been accepted for publication.
Access Criteria: Access to the data set will be limited to those persons who sign and submit a data use agreement that ensures protection of the confidentiality of the study participants.

REFERENCES:
- [Background] Pierce JS, Kozikowski C, Lee JM, Wysocki T. Type 1 diabetes in very young children: a model of parent and child influences on management and outcomes. Pediatr Diabetes. 2017 Feb;18(1):17-25. doi: 10.1111/pedi.12351. Epub 2015 Dec 29. PMID 26712357
- [Background] Pierce JS, Aroian K, Caldwell C, Ross JL, Lee JM, Schifano E, Novotny R, Tamayo A, Wysocki T. The Ups and Downs of Parenting Young Children With Type 1 Diabetes: A Crowdsourcing Study. J Pediatr Psychol. 2017 Sep 1;42(8):846-860. doi: 10.1093/jpepsy/jsx056. PMID 28369409
- [Background] Pierce JS, Wasserman R, Enlow P, Aroian K, Lee J, Wysocki T. Benefit finding among parents of young children with type 1 diabetes. Pediatr Diabetes. 2019 Aug;20(5):652-660. doi: 10.1111/pedi.12860. Epub 2019 May 20. PMID 31006941
- [Derived] Wilcocks CP, Enlow P, Wasserman R, Wysocki T, Lee J, Aroian K, Pierce JS. Development and Evaluation of the Pediatric Diabetes Routine Questionnaire for Parents of Young Children with Type 1 Diabetes. J Clin Psychol Med Settings. 2023 Mar;30(1):216-226. doi: 10.1007/s10880-022-09888-3. Epub 2022 Jun 18. PMID 35716238

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT03222180/Prot_SAP_001.pdf